CLINICAL TRIAL: NCT00808756
Title: Study on Fermentable Carbohydrates in Healthy Infants
Acronym: BAMBINOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Collaborators: Hospital Universitari Joan XXIII de Tarragona. (Other); Hospital Universitari Sant Joan (Unknown); Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Principal Investigator, Ricardo Closa-Monasterolo, Ricardo Closa Monasterolo, MD, PhD, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BAMBINOL
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Infant; Growth; Nutrition; Healthy
Keywords: Carbohydrates; Infant; Intestine; Faeces; Growth; Diet

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1: Intervention (Experimental): This group will be fed a diet enriched with fermentable carbohydrates.
  Interventions: Dietary Supplement: Fermentable carbohydrates.
- 2: Placebo. (Placebo Comparator): The placebo group will be fed a diet without addition of fermentable carbohydrates. This placebo formula will have the same nutritional values than the intervention (energy, proteins, carbohydrates, fat, vitamins & minerals).
  Interventions: Other: Standard infant formula.
- BF (No Intervention): The 2 intervention groups will be compared with a breast-fed infants control group.

INTERVENTIONS:
Dietary Supplement: Fermentable carbohydrates. — Infant formula enriched with fermentable carbohydrates.
  Arms: 1: Intervention
Other: Standard infant formula. — Standard infant formula.
  Arms: 2: Placebo.

SUMMARY:
The purpose of this project is to study the effect of fermentable carbohydrates in the nutrition of healthy infants.

DETAILED DESCRIPTION:
Breast-fed infants have a lower occurrence of episodes of sickness compared with formula-fed infants, and this has been ascribed to their different flora composition. The purpose of this project is to study the effect of fermentable carbohydrates in the nutrition of healthy infants. Additionally, other metabolic parameters will be investigated and compared to breast-fed infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants born in Reus and Tarragona area
* Healthy
* Normal feeding behaviour

Exclusion Criteria:

* Serious respiratory, neurological, gastrointestinal or metabolic disorders
* Infections or other serious diseases that could interfere in normal feeding or growth
* Parents or guardians cannot be expected to comply with protocol
* Parents or guardians have not command on Catalan or Spanish language

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 388 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Children well-being and appropriate growth | up to 4 months

SECONDARY OUTCOMES:
Secondary outcomes will be metabolic parameters. | Up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Closa, PhD, Prof, Principal Investigator — University Rovira i Virgili & Hospital Universitari Joan XXIII; Joaquin Escribano, PhD, Prof, Principal Investigator — Universitat Rovira i Virgili. Hospital Universitari Sant Joan de Reus.; Veronica Luque, PhD, Study Director — University Rovira i Virgili
Locations (2):
- Spain (2):
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona, Tarragona

REFERENCES:
- [Derived] Closa-Monasterolo R, Gispert-Llaurado M, Luque V, Ferre N, Rubio-Torrents C, Zaragoza-Jordana M, Escribano J. Safety and efficacy of inulin and oligofructose supplementation in infant formula: results from a randomized clinical trial. Clin Nutr. 2013 Dec;32(6):918-27. doi: 10.1016/j.clnu.2013.02.009. Epub 2013 Feb 26. PMID 23498848